CLINICAL TRIAL: NCT02755649
Title: A Phase 3 Study Investigating the Efficacy, Safety, and Tolerability of Dupilumab Administered to Adult Patients With Severe Atopic Dermatitis Who Are Not Adequately Controlled With or Are Intolerant to Oral Cyclosporine A, or When This Treatment is Not Medically Advisable
Brief Title: A Study to Assess the Efficacy and Safety of Dupilumab in Participants With Severe Atopic Dermatitis (AD) That Are Not Controlled With Oral Cyclosporine A (CSA) or for Those Who Cannot Take Oral CSA Because it is Not Medically Advisable
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R668-AD-1424
Record Dates: First submitted 2016-03-02; First posted 2016-04-29 (Estimated); Results first posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo QW + TCS (Experimental): Participants received one subcutaneous (SC) injection of dupilumab matching placebo once per week (QW) (following two SC injections on day 1) from Week 1 to Week 15. All participants were required to undergo treatment with topical corticosteroids (TCS) using a standardized regimen that continued through the end of the treatment period (Week 16). Starting at week 16, participants could roll over into an open-label extension (OLE) study (R668-AD-1225), if they were considered eligible. Participants who did not enter the OLE study were followed for up to an additional 12 weeks for safety ([Week 28, end of study (EOS) period]).
  Interventions: Drug: Matching Placebo
- Dupilumab 300 mg Q2W + TCS (Experimental): Participants received one subcutaneous (SC) injection of dupilumab 300 mg every 2 weeks (Q2W) from Week 1 to Week 15 (following a SC loading dose of 600 mg on day 1). During weeks in which dupilumab was not administered, participants received matching placebo. All participants were required to undergo treatment with topical corticosteroids (TCS) using a standardized regimen that continued through the end of the treatment period (Week 16). Starting at week 16, participants could roll over into an open-label extension (OLE) study (R668-AD-1225), if they were considered eligible. Participants who did not enter the OLE study were followed for up to an additional 12 weeks for safety ([Week 28, end of study (EOS) period]).
  Interventions: Drug: Dupilumab
- Dupilumab 300 mg QW + TCS (Experimental): Participants received one subcutaneous (SC) injection of dupilumab 300 mg once per week (QW) (following an SC loading dose of 600 mg on day 1) from Week 1 to Week 15. All participants were required to undergo treatment with topical corticosteroids (TCS) using a standardized regimen that continued through the end of the treatment period (Week 16). Starting at week 16, participants could roll over into an open-label extension (OLE) study (R668-AD-1225), if they were considered eligible. Participants who did not enter the OLE study were followed for up to an additional 12 weeks for safety ([Week 28, end of study (EOS) period]).
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab
  Other Names: DUPIXENT®; REGN668; SAR231893
  Arms: Dupilumab 300 mg Q2W + TCS; Dupilumab 300 mg QW + TCS
Drug: Matching Placebo
  Arms: Placebo QW + TCS

SUMMARY:
The main objective of the trial is to evaluate the efficacy of 2 dose regimens of dupilumab compared to placebo, administered with concomitant topical corticosteroids (TCS), in adult patients with severe AD who are not adequately controlled with, or are intolerant to, oral Cyclosporine A (CSA), or when this treatment is currently not medically advisable.

The secondary objective is to assess the safety and tolerability of 2 dose regimens of dupilumab compared to placebo, administered with concomitant TCS, in adult patients with severe AD who are not adequately controlled with, or are intolerant to, oral CSA, or when this treatment is currently not medically advisable.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years or older
2. Severe, Chronic AD, (according to American Academy of Dermatology Consensus Criteria [Eichenfield 2014]) for whom treatment with potent TCS is indicated
3. EASI score ≥20 at the screening and baseline visits
4. IGA score ≥3 (on the 0 to 4 IGA scale) at the screening and baseline visits
5. ≥10% body surface area (BSA) of AD involvement at the screening and baseline visits
6. Documented recent history (within 6 months before the screening visit) of inadequate response to treatment with TCS
7. Have applied a stable dose of topical emollient (moisturizer) twice daily for at least the 7 consecutive days immediately before the baseline visit
8. Documented history by a physician of either:

   1. No prior CSA exposure and not currently a candidate for CSA treatment due to:

      * medical contraindications (eg, uncontrolled hypertension on medication), or
      * use of prohibited concomitant medications (eg, statins, digoxin, macrolide, antibiotics, barbiturates, anti-seizure, nonsteroidal anti-inflammatory drugs, diuretics, angiotensin-converting-enzyme inhibitors, St John's Wort, etc), or
      * increased susceptibility to CSA-induced renal damage (elevated creatinine) and liver damage (elevated function tests), or
      * increased risk of serious infections, or
      * hypersensitivity to CSA active substance or excipients OR
   2. Previously exposed to CSA, and CSA treatment should not be continued or restarted due to:

      * intolerance and/or unacceptable toxicity (eg, elevated creatinine, elevated liver function tests, uncontrolled hypertension, paraesthesia, headache, nausea, hypertrichosis, etc), or
      * inadequate response to CSA (defined as flare of AD on CSA tapering after a maximum of 6 weeks of high dose [5 mg/kg/day] to maintenance dose [2 to 3 mg/kg/day] or a flare after a minimum of 3 months on maintenance dose). Flare is defined as increase in signs and/or symptoms leading to escalation of therapy, which can be an increase in dose, a switch to a higher-potency class of TCS, or the start of another systemic non-steroidal immunosuppressive drug or
      * requirement for CSA at doses >5 mg/kg/day, or duration beyond those specified in the prescribing information (>1 year)

Exclusion Criteria:

1. Participation in a prior dupilumab clinical study
2. Treatment with an investigational drug within 8 weeks or within 5 half-lives (if known), whichever is longer, before the screening visit
3. Hypersensitivity and/or intolerance to corticosteroids or to any other ingredients contained in the TCS product used in the study
4. Systemic CSA, systemic corticosteroids, or phototherapy within 4 weeks prior to screening, and azathioprine (AZA), methotrexate (MTX), mycophenolate mofetil (MMF), or Janus kinase (JAK) inhibitors within 8 weeks prior to screening
5. Treatment with TCI within 1 week before the screening visit
6. Treatment with biologics as follows:

   * Any cell-depleting agents including but not limited to rituximab: within 6 months before the screening visit, or until lymphocyte count returns to normal, whichever is longer
   * Other biologics: within 5 half-lives (if known) or 16 weeks prior to the screening visit, whichever is longer
7. Regular use (more than 2 visits per week) of a tanning booth/parlor within 4 weeks of the screening visit
8. Treatment with a live (attenuated) vaccine within 12 weeks before the screening
9. Active chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 2 weeks before the screening or superficial skin infections within 1 week before the screening visit. NOTE: patients may be rescreened no sooner than 2 weeks after infection resolves
10. Known or suspected history of immunosuppression, including history of invasive opportunistic infections (eg, tuberculosis [TB], histoplasmosis, Listeriosis, coccidioidomycosis, pneumocystosis, aspergillosis) despite infection resolution; or unusually frequent, recurrent, or prolonged infections, per investigator judgment
11. Presence of any 1 of the following TB criteria:

    1. A positive tuberculin skin test at the screening visit
    2. A positive blood QuantiFERON®-TB or T-Spot test at the screening visit
    3. Chest x-ray (posterior-anterior and lateral views) at screening or within 3 months before the screening visit (radiology report must be available) with results consistent with prior TB infection (including but not limited to apical scarring, apical fibrosis, or multiple calcified granuloma). This does not include non-caseating granulomata.

    NOTE: Any of these 3 TB tests will be performed on a country-by-country basis according to local guidelines only if required by regulatory authorities or ethics boards.
12. History of human immunodeficiency virus (HIV) infection or positive HIV serology at screening
13. Positive hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBc Ab), or hepatitis C antibody (HCV Ab) at the screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2016-01-31 (Actual); Primary Completion 2017-01-04 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (73):
- Austria (2):
  - Site 1, Vienna
  - Site 2, Vienna
- Belgium (3):
  - Brussels
  - Leuven
  - Loverval
- Germany (30):
  - Site 1, Berlin
  - Site 2, Berlin
  - Site 3, Berlin
  - Site 4, Berlin
  - Site 5, Berlin
  - Site 6, Berlin
  - Site 7, Berlin
  - Bochum
  - Site 1, Dresden
  - Site 2, Dresden
  - Site 3, Dresden
  - Erlangen
  - Frankfurt am Main
  - Site 1, Hamburg
  - Site 2, Hamburg
  - Heidelberg
  - Kiel
  - Langenau
  - Leipzig
  - Lübeck
  - Magdeburg
  - Mahlow
  - Mainz
  - Site 1, München
  - Site 2, München
  - Münster
  - Osnabrück
  - Selters
  - Stuttgart
  - Tübingen
- Dublin, Ireland
- Netherlands (2):
  - Amsterdam
  - Utrecht
- Poland (21):
  - Site 1, Bialystok
  - Site 1, Bydgoszcz
  - Site 2, Bydgoszcz
  - Gdansk
  - Site 1, Katowice
  - Site 2, Katowice
  - Site 3, Katowice
  - Kielce
  - Site 1, Krakow
  - Site 2, Krakow
  - Site 1, Lodz
  - Site 2, Lodz
  - Site 3, Lodz
  - Lublin
  - Szczecin
  - Site 1, Warsaw
  - Site 2, Warsaw
  - Warsaw
  - Site 1, Wroclaw
  - Site 2, Wroclaw
  - Zgierz
- Russia (5):
  - Chelyabinsk
  - Kazan'
  - Moscow
  - Ryazan
  - Saint Petersburg
- Slovakia (2):
  - Košice
  - Svidník
- Spain (2):
  - Site 1, Barcelona
  - Site 2, Barcelona
- United Kingdom (5):
  - Site 1, London
  - Site 2, London
  - Oxford
  - Portsmouth
  - Sheffield

REFERENCES:
- [Derived] Silverberg JI, Lynde CW, Abuabara K, Patruno C, de Benedetto A, Zhang H, Thomas RB, Bego-Le-Bagousse G, Khokhar FA, Vakil J, Marco AR, Levit NA. Efficacy and Safety of Dupilumab Maintained in Adults >/= 60 Years of Age with Moderate-to-Severe Atopic Dermatitis: Analysis of Pooled Data from Four Randomized Clinical Trials. Am J Clin Dermatol. 2023 May;24(3):469-483. doi: 10.1007/s40257-022-00754-4. Epub 2023 Feb 20. PMID 36808602
- [Derived] Paller AS, Silverberg JI, Cork MJ, Guttman-Yassky E, Lockshin B, Irvine AD, Kim MB, Kabashima K, Chen Z, Lu Y, Bansal A, Rossi AB, Shabbir A. Efficacy and Safety of Dupilumab in Patients With Erythrodermic Atopic Dermatitis: A Post Hoc Analysis of 6 Randomized Clinical Trials. JAMA Dermatol. 2023 Mar 1;159(3):255-266. doi: 10.1001/jamadermatol.2022.6192. PMID 36723913
- [Derived] Mickevicius T, Pink AE, Bhogal M, O'Brart D, Robbie SJ. Dupilumab-Induced, Tralokinumab-Induced, and Belantamab Mafodotin-Induced Adverse Ocular Events-Incidence, Etiology, and Management. Cornea. 2023 Apr 1;42(4):507-519. doi: 10.1097/ICO.0000000000003162. Epub 2022 Dec 15. PMID 36525340
- [Derived] Griffiths C, de Bruin-Weller M, Deleuran M, Fargnoli MC, Staumont-Salle D, Hong CH, Sanchez-Carazo J, Foley P, Seo SJ, Msihid J, Chen Z, Cyr SL, Rossi AB. Dupilumab in Adults with Moderate-to-Severe Atopic Dermatitis and Prior Use of Systemic Non-Steroidal Immunosuppressants: Analysis of Four Phase 3 Trials. Dermatol Ther (Heidelb). 2021 Aug;11(4):1357-1372. doi: 10.1007/s13555-021-00558-0. Epub 2021 Jun 18. PMID 34142350
- [Derived] Boguniewicz M, Beck LA, Sher L, Guttman-Yassky E, Thaci D, Blauvelt A, Worm M, Corren J, Soong W, Lio P, Rossi AB, Lu Y, Chao J, Eckert L, Gadkari A, Hultsch T, Ruddy M, Mannent LP, Graham NMH, Pirozzi G, Chen Z, Ardeleanu M. Dupilumab Improves Asthma and Sinonasal Outcomes in Adults with Moderate to Severe Atopic Dermatitis. J Allergy Clin Immunol Pract. 2021 Mar;9(3):1212-1223.e6. doi: 10.1016/j.jaip.2020.12.059. Epub 2021 Jan 13. PMID 33453450
- [Derived] Silverberg JI, Simpson EL, Guttman-Yassky E, Cork MJ, de Bruin-Weller M, Yosipovitch G, Eckert L, Chen Z, Ardeleanu M, Shumel B, Hultsch T, Rossi AB, Hamilton JD, Orengo JM, Ruddy M, Graham NMH, Pirozzi G, Gadkari A. Dupilumab Significantly Modulates Pain and Discomfort in Patients With Atopic Dermatitis: A Post Hoc Analysis of 5 Randomized Clinical Trials. Dermatitis. 2021 Oct 1;32(1S):S81-S91. doi: 10.1097/DER.0000000000000698. PMID 33165005
- [Derived] Eichenfield LF, Bieber T, Beck LA, Simpson EL, Thaci D, de Bruin-Weller M, Deleuran M, Silverberg JI, Ferrandiz C, Folster-Holst R, Chen Z, Graham NMH, Pirozzi G, Akinlade B, Yancopoulos GD, Ardeleanu M. Infections in Dupilumab Clinical Trials in Atopic Dermatitis: A Comprehensive Pooled Analysis. Am J Clin Dermatol. 2019 Jun;20(3):443-456. doi: 10.1007/s40257-019-00445-7. PMID 31066001
- [Derived] de Bruin-Weller M, Graham NMH, Pirozzi G, Shumel B. Could conjunctivitis in patients with atopic dermatitis treated with dupilumab be caused by colonization with Demodex and increased interleukin-17 levels?: reply from the authors. Br J Dermatol. 2018 May;178(5):1220-1221. doi: 10.1111/bjd.16348. Epub 2018 Mar 2. No abstract available. PMID 29336016

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 73 sites in Europe. A total of 390 participants were screened between 28 Jan 2016 and 14 Sep 2016. Of those, 325 participants were enrolled into the study and randomized. Sixty participants were considered screen failures, mostly due to unmet eligibility criteria.
Pre-assignment Details: After providing informed consent, participants were assessed for study eligibility. Screening assessments were performed between day -28 & day -15, prior to randomization. Participants who met eligibility criteria at baseline (day 1) were randomized in a 1:1:1 ratio to receive dupilumab (weekly [QW] or every 2 weeks [Q2W]) or placebo.
Groups:
- Placebo QW + TCS: Participants received one subcutaneous (SC) injection of matching placebo once per week (QW) (following two SC injections on day 1) from Week 1 to Week 15. All participants required to undergo treatment with topical corticosteroids (TCS) using standardized regimen that continued through the end of treatment period (Week 16). At week 16, participants could roll over into an open-label extension (OLE) study (R668-AD-1225), if considered eligible. Participants who did not enter the OLE study were followed for up to an additional 12 weeks for safety ([Week 28, end of study (EOS) period]).
Period: Overall Study
Arm/Group | Placebo QW + TCS | Dupilumab 300 mg Q2W + TCS | Dupilumab 300 mg QW + TCS
Started | 108 | 107 | 110
Completed Treatment (Week 16) | 107 | 106 | 109
Completed Study (Week 28) | 7 | 8 | 8
Completed | 7 | 8 | 8
Not Completed | 101 | 99 | 102
Not completed — Transitioned into OLE study | 99 | 98 | 100
Not completed — Did Not Complete Follow-up Visits | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Undecided | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo QW + TCS | Dupilumab 300 mg Q2W + TCS | Dupilumab 300 mg QW + TCS | Total
Number analyzed (Participants) | 108 | 107 | 110 | 325
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (13.35) | 37.5 (12.89) | 38.7 (13.21) | 38.4 (13.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 42 | 44 | 126
  Male | 68 | 65 | 66 | 199
Eczema Area and Severity Index (EASI) Score [Mean (Standard Deviation); unit: Score on a Scale] — The EASI score is used to measure the severity and extent of atopic dermatitis (AD) and measured erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD.
  Score on a Scale | 32.9 (10.80) | 33.3 (9.93) | 33.1 (11.02) | 33.1 (10.56)
Peak Weekly Averaged Pruritus Numerical Rating Scale (NRS) score [Mean (Standard Deviation); unit: Score on a Scale] — Pruritus NRS is an assessment tool used to report intensity of participant's pruritus (itch), both average & maximum intensity, during 24-hr recall period. Participants were asked two questions: 1) For average itch intensity: how would you rate your itch overall (on average) during the previous 24 hrs; & 2) For maximum itch intensity: How would you rate your itch at the worst moment during the previous 24 hrs? Both questions were rated on a scale: 0-10 with 0=no itch & 10=worst itch imaginable. Population: Here "Number of Participants Analyzed" = Participants who were evaluable for this baseline characteristic
  Score on a Scale
    number analyzed (Participants) | 107 | 107 | 110 | 324
    (all) | 6.4 (2.23) | 6.6 (2.10) | 6.2 (2.01) | 6.4 (2.11)
Body Surface Area (BSA) Involvement of Atopic Dermatitis [Mean (Standard Deviation); unit: Score on a Scale] — BSA affected by AD was assessed for each section of the body (the possible highest score for each region was: head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%]). It was reported as a percentage of all major body sections combined.
  Score on a Scale | 55.0 (20.51) | 56.1 (17.83) | 56.0 (19.26) | 55.7 (19.18)
Global Individual Signs Score (GISS) [Mean (Standard Deviation); unit: Score on a Scale] — Individual components of the AD lesions (erythema, infiltration/papulation, excoriations, and lichenification) were rated globally (each assessed for the whole body, not by anatomical region) on a 4-point scale (0 = none, 1 = mild, 2 = moderate and 3 = severe) using the EASI severity grading criteria. Total score ranges from 0 (absent disease) to 12 (severe disease).
  Score on a Scale | 9.4 (1.63) | 9.3 (1.64) | 9.1 (1.63) | 9.3 (1.64)
Dermatology Life Quality Index (DLQI) Total Score [Mean (Standard Deviation); unit: Score on a Scale] — The DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on quality of life (QOL). The 10 questions assessed QOL over the past week, with individual scoring per question of 0 (not at all) to 3 (very much) and an overall scoring of 0 (absent disease) to 30 (severe disease); a high score indicative of a poor QOL.
  Score on a Scale | 13.2 (7.60) | 14.5 (7.63) | 13.8 (8.03) | 13.8 (7.75)
Patient Oriented Eczema Measure (POEM) [Mean (Standard Deviation); unit: Score on a Scale] — The POEM is a 7-item questionnaire that assessed disease symptoms (dryness, itching, flaking, cracking, sleep loss, bleeding and weeping) with a scoring system of 0 (absent disease) to 28 (severe disease) (high score indicative of poor QOL) Population: Here "Number of Participants Analyzed" = Participants who were evaluable for this baseline characteristic
  Score on a Scale
    number analyzed (Participants) | 107 | 107 | 110 | 324
    (all) | 19.1 (5.99) | 19.3 (6.21) | 18.6 (6.97) | 19.0 (6.40)
Total Hospital Anxiety and Depression Scale (HADS) [Mean (Standard Deviation); unit: Score on a Scale] — The HADS is a 14-item scale, with 7 items relating to anxiety and 7 relating to depression. Each item on the questionnaire is scored from 0-3, for possible scores ranging from 0 (no symptoms) to 21 (severe symptoms) for each of the anxiety and depression subscales. Recommended cut-off scores for both subscales to identify psychiatric distress are: 7 to 8 for possible presence, 10 to 11 for probable presence, and 14 to 15 for severe anxiety or depression. Scores less than 7 do not indicate psychiatric distress. Total score is the sum of the two sub-scores.
  Score on a Scale | 13.0 (7.85) | 12.8 (8.01) | 13.3 (8.15) | 13.0 (7.98)
SCORing Atopic Dermatitis (SCORAD) score [Mean (Standard Deviation); unit: Score on a Scale] — The SCORAD is a clinical tool for assessing the extent and severity of AD. Extent and intensity of eczema as well as subjective symptoms (insomnia, etc.) were assessed and scored. Total score ranges from 0 (absent disease) to 103 (severe disease).
  Score on a Scale | 67.0 (12.20) | 68.6 (11.91) | 66.0 (12.70) | 67.2 (12.29)
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 5 | 9
  Not Hispanic or Latino | 101 | 99 | 101 | 301
  Not Reported/Missing | 4 | 7 | 4 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  White | 104 | 104 | 105 | 313
  Black or African American | 0 | 0 | 2 | 2
  Asian | 2 | 2 | 2 | 6
  Other | 2 | 0 | 1 | 3
  Not Reported / Missing | 0 | 1 | 0 | 1
Investigator's Global Assessment (IGA) score [Count of Participants; unit: Participants] — IGA is an assessment scale used to determine severity of AD and clinical response to treatment on a 5-point scale (0 = clear; 1= almost clear; 2= mild; 3= moderate; 4= severe) based on erythema and papulation/ infiltration. Therapeutic response is an IGA score of 0 (clear) or 1 (almost clear).
  Participants
    IGA score = 3 | 56 | 57 | 58 | 171
    IGA score = 4 | 52 | 50 | 52 | 154

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Eczema Area and Severity Index (EASI) 75 (≥75% Improvement From Baseline) at Week 16
Description: The EASI score is used to measure the severity and extent of atopic dermatitis (AD) and measured erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. EASI-75 responders were the participants who achieved ≥75% overall improvement in EASI score from baseline to Week 16. The analysis population for efficacy analyses is the Full Analysis Set (FAS) which included all randomized participants. Efficacy analyses were based on the treatment allocated (as randomized).
Time Frame: Baseline, Week 16
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo QW + TCS | Dupilumab 300 mg Q2W + TCS | Dupilumab 300 mg QW + TCS
Number analyzed (Participants) | 108 | 107 | 110
Percentage of Participants | 29.6 | 62.6 | 59.1
Statistical Analysis 1: Comparison: Placebo QW + TCS vs Dupilumab 300 mg QW + TCS; A hierarchical testing approach was used to control Type-1 error at 0.05 across 2 dose regimens. Difference is Dupilumab minus placebo. Confidence Interval (CI) calculated using normal approximation. Participants with missing values at Week 16 were categorized as non-responders at Week 16. Participants who used rescue treatment were categorized as non-responders from time rescue treatment was initiated; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level. P-values were derived by Cochran-Mantel-Haenszel (CMH) test stratified by disease severity (IGA 3 vs IGA 4) and prior Cyclosporine A (CSA) use (Yes, No); Difference in Percentages = 29.5, 95% CI 2-sided [16.87 to 42.05]
Statistical Analysis 2: Comparison: Placebo QW + TCS vs Dupilumab 300 mg Q2W + TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; difference in percentages = 33, 95% CI 2-sided [20.41 to 45.57]

2. Secondary Outcome: Percent Change From Baseline in Eczema Area and Severity Index (EASI) Score at Week 16
Description: The EASI score is used to measure the severity and extent of atopic dermatitis (AD) and measured erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. The analysis population for efficacy analyses is the FAS which included all randomized participants. Efficacy analyses were based on the treatment allocated (as randomized). Here "number of participants analyzed" = participants who were evaluable for this endpoint.
Time Frame: Baseline, Week 16
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo QW + TCS | Dupilumab 300 mg Q2W + TCS | Dupilumab 300 mg QW + TCS
Number analyzed (Participants) | 89 | 103 | 105
Percent Change | -46.6 (2.76) [lower limit 2.76] | -79.8 (2.59) [lower limit 2.59] | -78.2 (2.55) [lower limit 2.55]
Statistical Analysis 1: Comparison: Placebo QW + TCS vs Dupilumab 300 mg QW + TCS; Hierarchical testing approach to control Type-1 error rate at 0.05 across 2 dose regimens.CI w/p-value based on treatment difference(dupilumab vs placebo) of LS mean percent change using multiple imputation (MI) w/ANCOVA model w/baseline measurement as covariate & treatment, randomization strata(disease severity[IGA 3 vs IGA 4] & prior CSA use[Yes,No]) as fixed factors.Efficacy data from participants who received rescue treatment were set to missing after timepoint of rescue, then imputed by MI; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; Least square (LS) mean difference = -31.6, 95% CI 2-sided [-38.85 to -24.3]
Statistical Analysis 2: Comparison: Placebo QW + TCS vs Dupilumab 300 mg Q2W + TCS; Hierarchical testing approach was used to control Type-1 error rate at 0.05 across 2 dose regimens.CI with p-value based on treatment difference(dupilumab vs. placebo) of LS mean percent change using MI with ANCOVA model with baseline measurement as covariate & treatment, randomization strata(disease severity[IGA 3 vs IGA 4] & prior CSA use [Yes,No]) as fixed factors. Efficacy data from participants who received rescue treatment were set to missing after timepoint of rescue & then imputed by MI; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -33.1, 95% CI 2-sided [-40.42 to -25.88]

3. Secondary Outcome: Percent Change From Baseline in Weekly Average of Peak Pruritus Numerical Rating Scale (NRS) at Week 16
Description: The Pruritus NRS is an assessment tool used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would you rate your itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). The analysis population for efficacy analyses is the FAS. Efficacy analyses were based on the treatment allocated (as randomized). Here "Number of Participants Analyzed" = Participants who were evaluable for this endpoint.
Time Frame: Baseline, Week 16
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo QW + TCS | Dupilumab 300 mg Q2W + TCS | Dupilumab 300 mg QW + TCS
Number analyzed (Participants) | 89 | 102 | 103
Percent Change | -25.4 (3.39) | -53.9 (3.14) | -51.7 (3.09)
Statistical Analysis 1: Comparison: Placebo QW + TCS vs Dupilumab 300 mg QW + TCS; Hierarchical testing approach was used to control Type-1 error rate at 0.05 across 2 dose regimens.CI with p-value based on treatment difference(dupilumab vs. placebo) of LS mean percent change using MI with ANCOVA model with baseline measurement as covariate & treatment, randomization strata(disease severity[IGA 3 vs IGA 4] & prior CSA use [Yes,No]) as fixed factors.Efficacy data from participants who received rescue treatment were set to missing after timepoint of rescue, then imputed by MI; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS mean difference = -26.2, 95% CI 2-sided [-35.07 to -17.41]
Statistical Analysis 2: Comparison: Placebo QW + TCS vs Dupilumab 300 mg Q2W + TCS; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference] = -28.5, 95% CI 2-sided [-37.34 to -19.68]

4. Secondary Outcome: Percent Change From Baseline in SCORing Atopic Dermatitis (SCORAD) Score at Week 16
Description: The SCORAD is a clinical tool for assessing the severity of AD. Extent and intensity of eczema as well as subjective signs (insomnia, etc.) are assessed and scored. Total score ranges from 0 (absent disease) to 103 (severe disease). The analysis population for efficacy analyses is the FAS. Efficacy analyses were based on the treatment allocated (as randomized). Here "Number of Participants analyzed" = Participants who were evaluable for this endpoint.
Time Frame: Baseline, Week 16
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo QW + TCS | Dupilumab 300 mg Q2W + TCS | Dupilumab 300 mg QW + TCS
Number analyzed (Participants) | 89 | 103 | 104
Percent Change | -29.5 (2.55) [lower limit 2.55] | -62.4 (2.48) [lower limit 2.48] | -58.3 (2.45) [lower limit 2.45]
Statistical Analysis 1: Comparison: Placebo QW + TCS vs Dupilumab 300 mg QW + TCS; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -28.7, 95% CI 2-sided [-35.56 to -21.93]
Statistical Analysis 2: Comparison: Placebo QW + TCS vs Dupilumab 300 mg Q2W + TCS; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -32.9, 95% CI 2-sided [-39.7 to -26.06]

5. Secondary Outcome: Percentage of Participants With Improvement (Reduction ≥4 Points) of Weekly Average of Peak Daily Pruritus NRS From Baseline to Week 16
Description: Pruritus NRS is an assessment tool used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). Participants achieving a reduction of ≥4 points from baseline in weekly average of peak daily pruritus NRS score at Week 16 were reported. The analysis population for efficacy analyses is the FAS. Efficacy analyses were based on the treatment allocated (as randomized). Here "Number of participants analyzed" = participants who were evaluable for this endpoint.
Time Frame: Baseline to Week 16
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo QW + TCS | Dupilumab 300 mg Q2W + TCS | Dupilumab 300 mg QW + TCS
Number analyzed (Participants) | 91 | 94 | 94
Percentage of participants | 14.3 | 45.7 | 40.4
Statistical Analysis 1: Comparison: Placebo QW + TCS vs Dupilumab 300 mg QW + TCS; A hierarchical testing approach was used to control Type-1 error at 0.05 across the 2 dose regimens. Difference is dupilumab minus placebo. CI calculated using normal approximation. P-values were derived by CMH test stratified by disease severity (IGA 3 vs IGA 4) and prior CSA use (Yes,No). Participants who used rescue treatment were categorized as non-responders from time rescue treatment was initiated. Participants with missing values at Week 16 were categorized as non-responders at Week 16; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; difference in percentages = 26.1, 95% CI 2-sided [13.89 to 38.39]
Statistical Analysis 2: Comparison: Placebo QW + TCS vs Dupilumab 300 mg Q2W + TCS; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; difference in percentages = 31.5, 95% CI 2-sided [19.08 to 43.83]

6. Secondary Outcome: Change From Baseline in Percent Body Surface Area (BSA) Involvement With Atopic Dermatitis (AD) at Week 16
Description: BSA affected by AD was assessed for each section of the body (the possible highest score for each region was: head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%]). It was reported as a percentage of all major body sections combined. The analysis population for efficacy analyses is the FAS. Efficacy analyses were based on the treatment allocated (as randomized). Here "number of participants analyzed" = participants who were evaluable for this endpoint.
Time Frame: Baseline, Week 16
Measure: Least Squares Mean (Standard Error); unit: Percent BSA
Arm/Group | Placebo QW + TCS | Dupilumab 300 mg Q2W + TCS | Dupilumab 300 mg QW + TCS
Number analyzed (Participants) | 89 | 103 | 104
Percent BSA | -19.57 (1.798) [lower limit 1.798] | -39.23 (1.715) [lower limit 1.715] | -37.52 (1.690) [lower limit 1.690]
Statistical Analysis 1: Comparison: Placebo QW + TCS vs Dupilumab 300 mg QW + TCS; Hierarchical testing approach was used to control Type-1 error rate at 0.05 across 2 dose regimens.CI with p-value is based on treatment difference(dupilumab vs. placebo) of LS mean percent change using MI with ANCOVA model with baseline measurement as covariate & treatment,randomization strata(disease severity[IGA 3 vs IGA 4] & prior CSA use [Yes,No]) as fixed factors. Efficacy data from participants who received rescue treatment were set to missing after timepoint of rescue, then imputed by MI; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -17.95, 95% CI 2-sided [-22.706 to -13.197]
Statistical Analysis 2: Comparison: Placebo QW + TCS vs Dupilumab 300 mg Q2W + TCS; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -19.66, 95% CI 2-sided [-24.431 to -14.895]

7. Secondary Outcome: Percentage of Participants With Investigator Global Assessment (IGA) 0 or 1 (on the 0 to 4 IGA Scale) and a Reduction From Baseline of ≥2 Points at Week 16
Description: IGA is an assessment scale used to determine severity of AD and clinical response to treatment on a 5 point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic response is an IGA score of 0 (clear) or 1 (almost clear). Participants with IGA score of "0" or "1" and a reduction from baseline of ≥2 points at Week 16 were reported. The analysis population for efficacy analyses is the FAS. Efficacy analyses were based on the treatment allocated (as randomized).
Time Frame: Baseline, Week 16
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo QW + TCS | Dupilumab 300 mg Q2W + TCS | Dupilumab 300 mg QW + TCS
Number analyzed (Participants) | 108 | 107 | 110
Percentage of Participants | 13.9 | 40.2 | 39.1
Statistical Analysis 1: Comparison: Placebo QW + TCS vs Dupilumab 300 mg QW + TCS; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Difference in Percentages = 25.2, 95% CI 2-sided [13.99 to 36.41]
Statistical Analysis 2: Comparison: Placebo QW + TCS vs Dupilumab 300 mg Q2W + TCS; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Difference in Percentages = 26.3, 95% CI 2-sided [14.95 to 37.65]

8. Secondary Outcome: Change From Baseline in the Dermatology Life Quality Index (DLQI) at Week 16
Description: The DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on quality of life (QOL). The 10 questions assessed QOL over the past week, with an overall scoring of 0 (absent disease) to 30 (severe disease); a high score is indicative of a poor QOL. The analysis population for efficacy analyses is the FAS. Efficacy analyses were based on the treatment allocated (as randomized). Here "Number of Participants Analyzed" = Participants who were evaluable for this endpoint.
Time Frame: Baseline, Week 16
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo QW + TCS | Dupilumab 300 mg Q2W + TCS | Dupilumab 300 mg QW + TCS
Number analyzed (Participants) | 89 | 103 | 104
Score on a Scale | -4.5 (0.49) [lower limit 0.49] | -9.5 (0.46) [lower limit 0.46] | -8.8 (0.45) [lower limit 0.45]
Statistical Analysis 1: Comparison: Placebo QW + TCS vs Dupilumab 300 mg QW + TCS; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -4.3, 95% CI 2-sided [-5.6 to -3.04]
Statistical Analysis 2: Comparison: Placebo QW + TCS vs Dupilumab 300 mg Q2W + TCS; Hierarchical testing approach was used to control Type-1 error rate at 0.05 across 2 dose regimens.CI with p-value based on treatment difference(dupilumab vs. placebo) of LS mean percent change using MI with ANCOVA model with baseline measurement as covariate & treatment, randomization strata(disease severity[IGA 3 vs IGA 4] & prior CSA use [Yes,No])as fixed factors. Efficacy data from participants who received rescue treatment were set to missing after timepoint of rescue, then imputed by MI; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -5, 95% CI 2-sided [-6.31 to -3.74]

9. Secondary Outcome: Change From Baseline in the Patient Oriented Eczema Measure (POEM) at Week 16
Description: The POEM is a 7-item questionnaire that assesses disease symptoms (dryness, itching, flaking, cracking, sleep loss, bleeding and weeping) with a scoring system of 0 (absent disease) to 28 (severe disease) (high score indicative of poor quality of life [QOL]). The analysis population for efficacy analyses is the FAS. Efficacy analyses were based on the treatment allocated (as randomized). Here "Number of Participants Analyzed" = participants who were evaluable for this endpoint.
Time Frame: Baseline, Week 16
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo QW + TCS | Dupilumab 300 mg Q2W + TCS | Dupilumab 300 mg QW + TCS
Number analyzed (Participants) | 88 | 103 | 104
Score on a Scale | -4.3 (0.62) [lower limit 0.62] | -11.9 (0.60) [lower limit 0.60] | -11.4 (0.59) [lower limit 0.59]
Statistical Analysis 1: Comparison: Placebo QW + TCS vs Dupilumab 300 mg QW + TCS; [analysis description as in outcome 8, analysis 2]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -7.1, 95% CI 2-sided [-8.78 to -5.47]
Statistical Analysis 2: Comparison: Placebo QW + TCS vs Dupilumab 300 mg Q2W + TCS; [analysis description as in outcome 8, analysis 2]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -7.6, 95% CI 2-sided [-9.29 to -5.97]

10. Secondary Outcome: Percentage of Participants With Eczema Area and Severity Index (EASI) Score (≥75% Improvement From Baseline) at Week 16 for Participants With Prior CSA Use
Description: The EASI score is used to measure the severity and extent of atopic dermatitis (AD) and measured erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. EASI-75 responders were the participants who achieved ≥75% overall improvement in EASI score from baseline to Week 16. The analysis population for efficacy analyses is the FAS. Efficacy analyses were based on the treatment allocated (as randomized). Here "Number of Participants Analyzed" = Participants who were evaluable for this endpoint.
Time Frame: Baseline, Week 16
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo QW + TCS | Dupilumab 300 mg Q2W + TCS | Dupilumab 300 mg QW + TCS
Number analyzed (Participants) | 72 | 69 | 69
Percentage of Participants | 26.4 | 58.0 | 56.5
Statistical Analysis 1: Comparison: Placebo QW + TCS vs Dupilumab 300 mg QW + TCS; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Difference in Percentages = 30.1, 95% CI 2-sided [14.63 to 45.64]
Statistical Analysis 2: Comparison: Placebo QW + TCS vs Dupilumab 300 mg Q2W + TCS; Hierarchical testing approach was used to control Type-1 error at 0.05 across the 2 dose regimens. Difference is dupilumab minus placebo. CI calculated using normal approximation. P-values derived by CMH test stratified by disease severity (IGA 3 vs IGA 4) and prior CSA use (Yes,No). Participants who used rescue treatment were categorized as non-responders from time rescue treatment was initiated. Participants with missing values at Week 16 were categorized as non-responders at Week 16; Test type: Superiority; p = 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Difference in Percentages = 31.6, 95% CI 2-sided [16.11 to 47.05]

11. Secondary Outcome: Change From Baseline in Mean Weekly Dose of Topical Corticosteroid (TCS) Use During Treatment Period
Description: The type, amount, frequency, and potency of topical products used during the study were recorded at home by participants in a medication diary. Participants returned TCS tubes at each clinic visit up until week 16, and these tubes were weighed by the site staff to determine the actual amount of TCS used. During the 16-week placebo-controlled study treatment period, medium-potency TCS dosing frequency was symptom-based (IGA score) adjusted every 4 weeks per the protocol-specified tapering algorithm. The analysis population for efficacy analyses is the FAS. Efficacy analyses were based on the treatment allocated (as randomized). Here "Number Analyzed" = Participants who were evaluable for this endpoint.
Time Frame: Baseline to week 16
Measure: Least Squares Mean (Standard Error); unit: Grams
Arm/Group | Placebo QW + TCS | Dupilumab 300 mg Q2W + TCS | Dupilumab 300 mg QW + TCS
Number analyzed (Participants) | 108 | 107 | 110
Grams | 25.1 (1.48) [lower limit 1.48] | 15.0 (1.51) [lower limit 1.51] | 17.5 (1.49) [lower limit 1.49]
Statistical Analysis 1: Comparison: Placebo QW + TCS vs Dupilumab 300 mg QW + TCS; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0003, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -7.6, 95% CI 2-sided [-11.64 to -3.51]
Statistical Analysis 2: Comparison: Placebo QW + TCS vs Dupilumab 300 mg QW + TCS; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -10.1, 95% CI 2-sided [-14.15 to -5.95]

12. Secondary Outcome: Change From Baseline in Total Hospital Anxiety and Depression Scale (HADS) Score at Week 16
Description: The HADS is a 14-item scale, with 7 items relating to anxiety and 7 relating to depression. Each item on the questionnaire is scored from 0-3, for possible scores ranging from 0 (no symptoms) to 21 (severe symptoms) for each of the anxiety and depression subscales. Recommended cut-off scores for both subscales to identify psychiatric distress are: 7 to 8 for possible presence, 10 to 11 for probable presence, and 14 to 15 for severe anxiety or depression. Scores less than 7 do not indicate psychiatric distress. Total score is the sum of the two sub-scores.
Time Frame: Baseline, Week 16
Population: Analysis population for efficacy analyses is the FAS. Efficacy analyses were based on the treatment allocated (as randomized). Here "Number of Participants Analyzed" = Participants who were evaluable for this endpoint.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo QW + TCS | Dupilumab 300 mg Q2W + TCS | Dupilumab 300 mg QW + TCS
Number analyzed (Participants) | 89 | 103 | 104
Score on a Scale | -2.3 (0.56) [lower limit 0.56] | -6.1 (0.54) [lower limit 0.54] | -5.2 (0.53) [lower limit 0.53]
Statistical Analysis 1: Comparison: Placebo QW + TCS vs Dupilumab 300 mg QW + TCS; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -2.9, 95% CI 2-sided [-4.41 to -1.43]
Statistical Analysis 2: Comparison: Placebo QW + TCS vs Dupilumab 300 mg Q2W + TCS; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -3.9, 95% CI 2-sided [-5.38 to -2.4]

13. Secondary Outcome: Percentage of Participants Achieving SCORAD 50 (≥50% Improvement From Baseline) at Week 16
Description: The SCORAD is a clinical tool for assessing the severity of AD. Extent and intensity of eczema as well as subjective signs (insomnia, etc.) are assessed and scored. Total score ranges from 0 (absent disease) to 103 (severe disease). The analysis population for efficacy analyses is the FAS. Efficacy analyses were based on the treatment allocated (as randomized).
Time Frame: Baseline, Week 16
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo QW + TCS | Dupilumab 300 mg Q2W + TCS | Dupilumab 300 mg QW + TCS
Number analyzed (Participants) | 108 | 107 | 110
Percentage of Participants | 25.9 | 66.4 | 55.5
Statistical Analysis 1: Comparison: Placebo QW + TCS vs Dupilumab 300 mg QW + TCS; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Difference in Percentages = 29.5, 95% CI 2-sided [17.1 to 41.96]
Statistical Analysis 2: Comparison: Placebo QW + TCS vs Dupilumab 300 mg Q2W + TCS; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Difference in Percentages = 40.4, 95% CI 2-sided [28.24 to 52.61]

14. Secondary Outcome: Percent Change From Baseline in the Total Global Individual Signs Score (GISS) at Week 16 (Erythema, Infiltration/ Papulation, Excoriations, Lichenification)
Description: Individual components of the AD lesions (erythema, infiltration/ papulation, excoriations, and lichenification) were rated globally (each assessed for the whole body, not by anatomical region) on a 4-point scale (0= none, 1= mild, 2= moderate and 3= severe) using the EASI severity grading criteria. Total score ranges from 0 (absent disease) to 12 (severe disease). The analysis population for efficacy analyses is the FAS. Efficacy analyses were based on the treatment allocated (as randomized). Full Analysis Set (FAS) included all randomized. Here "Number of Participants Analyzed" = Participants who were evaluable for this endpoint.
Time Frame: Baseline, Week 16
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo QW + TCS | Dupilumab 300 mg Q2W + TCS | Dupilumab 300 mg QW + TCS
Number analyzed (Participants) | 89 | 103 | 104
Percent Change | -29.0 (2.75) [lower limit 2.75] | -55.2 (2.66) [lower limit 2.66] | -53.3 (2.65) [lower limit 2.65]
Statistical Analysis 1: Comparison: Placebo QW + TCS vs Dupilumab 300 mg QW + TCS; A hierarchical testing approach was used to control Type-1 error rate at 0.05 across 2 dose regimens.CI with p-value based on treatment difference(dupilumab group vs. placebo)of LS mean percent change using MI with ANCOVA with baseline measurement as covariate & treatment,randomization strata(disease severity[IGA 3 vs IGA 4] & prior CSA use[Yes,No])as fixed factors.Efficacy data from participants who received rescue treatment were set to missing after timepoint of rescue, then imputed by MI; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -24.3, 95% CI 2-sided [-31.63 to -16.88]
Statistical Analysis 2: Comparison: Placebo QW + TCS vs Dupilumab 300 mg Q2W + TCS; Hierarchical testing approach was used to control Type-1 error rate at 0.05 across 2 dose regimens.CI with p-value based on treatment difference(dupilumab vs. placebo) of LS mean percent change using MI with ANCOVA model with baseline measurement as covariate & treatment, randomization strata (disease severity[IGA 3 vs IGA 4] & prior CSA use [Yes,No]) as fixed factors.Efficacy data from participants who received rescue treatment were set to missing after timepoint of rescue, then imputed by MI; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -26.2, 95% CI 2-sided [-33.49 to -18.86]

15. Secondary Outcome: Percent Change From Baseline in Weekly Average of Peak Pruritus Numerical Rating Scale (NRS) Score at Week 2
Description: Pruritus NRS is an assessment tool used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would you rate your itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). The analysis population for efficacy analyses is the FAS. Efficacy analyses were based on the treatment allocated (as randomized). Here "Number of Participants analyzed" = Participants who were evaluable for this endpoint.
Time Frame: Baseline, Week 2
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo QW + TCS | Dupilumab 300 mg Q2W + TCS | Dupilumab 300 mg QW + TCS
Number analyzed (Participants) | 105 | 105 | 110
Percent Change | -10.0 (2.24) [lower limit 2.24] | -17.2 (2.25) [lower limit 2.25] | -19.7 (2.21) [lower limit 2.21]
Statistical Analysis 1: Comparison: Placebo QW + TCS vs Dupilumab 300 mg QW + TCS; Hierarchical testing approach was used to control Type-1 error rate at 0.05 across 2 dose regimens. CI with p-value based on treatment difference(dupilumab vs. placebo) of LS mean percent change using MI with ANCOVA model with baseline measurement as covariate & treatment, randomization strata(disease severity[IGA 3 vs IGA 4] & prior CSA use [Yes,No]) as fixed factors.Efficacy data from participants who received rescue treatment were set to missing after timepoint of rescue, then imputed by MI; Test type: Superiority; p = 0.0017, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -9.7, 95% CI 2-sided [-15.8 to -3.66]
Statistical Analysis 2: Comparison: Placebo QW + TCS vs Dupilumab 300 mg Q2W + TCS; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0214, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -7.2, 95% CI 2-sided [-13.31 to -1.06]

16. Secondary Outcome: Percentage of Participants With Skin Infection Treatment Emergent Adverse Events (TEAEs) (Excluding Herpetic Infections) From Baseline Through Treatment Period
Description: Treatment-emergent adverse events (TEAEs) were defined as AEs that developed or worsened or became serious during on-treatment period (time from the first dose of study drug to the last study dose (Week 16). A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. Any TEAE included participants with both serious and non-serious AEs. Safety analysis set (SAF) included all randomized participants who received any study drug; it was based on the treatment received (as treated).
Time Frame: Baseline to Week 16
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo QW + TCS | Dupilumab 300 mg Q2W + TCS | Dupilumab 300 mg QW + TCS
Number analyzed (Participants) | 108 | 107 | 110
Percentage of Participants | 8.3 | 1.9 | 3.6
Statistical Analysis 1: Comparison: Placebo QW + TCS vs Dupilumab 300 mg QW + TCS; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.1486, Cochran-Mantel-Haenszel; Difference in Percentages = -4.7, 95% CI 2-sided [-10.97 to 1.58]
Statistical Analysis 2: Comparison: Placebo QW + TCS vs Dupilumab 300 mg Q2W + TCS; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0319, Cochran-Mantel-Haenszel; Difference in Percentages = -6.5, 95% CI 2-sided [-12.27 to -0.65]

17. Secondary Outcome: Percentage of Participants Having at Least One Serious Treatment Emergent Adverse Event (TEAE) Through Treatment Period
Description: Treatment-emergent adverse events (TEAEs) were defined as AEs that developed or worsened or became serious during on-treatment period (time from the first dose of study drug to the last study dose (Week 16). A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. Any TEAE included participants with both serious and non-serious AEs. SAF included all randomized participants who received any study drug; it was based on the treatment received (as treated).
Time Frame: Baseline to Week 16
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo QW + TCS | Dupilumab 300 mg Q2W + TCS | Dupilumab 300 mg QW + TCS
Number analyzed (Participants) | 108 | 107 | 110
Percentage of Participants | 1.9 | 1.9 | 1.8
Statistical Analysis 1: Comparison: Placebo QW + TCS vs Dupilumab 300 mg QW + TCS; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.9829, Cochran-Mantel-Haenszel; difference in percentages = 0, 95% CI 2-sided [-3.6 to 3.53]
Statistical Analysis 2: Comparison: Placebo QW + TCS vs Dupilumab 300 mg Q2W + TCS; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 1, Cochran-Mantel-Haenszel; difference in percentages = 0, 95% CI 2-sided [-3.6 to 3.63]

18. Secondary Outcome: Percentage of Participants Having at Least One Treatment-Emergent Adverse Event (TEAE) Leading to Treatment Discontinuation Through Treatment Period
Description: as for outcome 17
Time Frame: Baseline to Week 16
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo QW + TCS | Dupilumab 300 mg Q2W + TCS | Dupilumab 300 mg QW + TCS
Number analyzed (Participants) | 108 | 107 | 110
Percentage of participants | 0.9 | 0 | 1.8
Statistical Analysis 1: Comparison: Placebo QW + TCS vs Dupilumab 300 mg QW + TCS; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.5619, Cochran-Mantel-Haenszel; difference in percentages = 0.9, 95% CI 2-sided [-2.19 to 3.97]
Statistical Analysis 2: Comparison: Placebo QW + TCS vs Dupilumab 300 mg Q2W + TCS; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.3241, Cochran-Mantel-Haenszel; difference in percentages = -0.9, 95% CI 2-sided [-2.73 to 0.88]

19. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events Through Treatment Period
Description: as for outcome 17
Time Frame: Baseline to Week 16
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo QW + TCS | Dupilumab 300 mg Q2W + TCS | Dupilumab 300 mg QW + TCS
Number analyzed (Participants) | 108 | 107 | 110
Percentage of participants | 69.4 | 72.0 | 69.1
Statistical Analysis 1: Comparison: Placebo QW + TCS vs Dupilumab 300 mg QW + TCS; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.9518, Cochran-Mantel-Haenszel; difference in percentages = -0.4, 95% CI 2-sided [-12.6 to 11.9]
Statistical Analysis 2: Comparison: Placebo QW + TCS vs Dupilumab 300 mg Q2W + TCS; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.6833, Cochran-Mantel-Haenszel; difference in percentages = 2.5, 95% CI 2-sided [-9.64 to 14.68]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of informed consent form up to end of study (EOS), Week 28, regardless of seriousness or relationship to investigational product.
Description: Pre-treatment AEs were AEs that developed/worsened in severity during pre-treatment period (from informed consent to first dose of study drug); All AEs collected during treatment and follow-up period were considered treatment emergent AEs (TEAEs). TEAEs were AEs that developed or worsened in severity compared to baseline during treatment and follow-up period.
Arm/Group | Placebo QW + TCS | Dupilumab 300 mg Q2W + TCS | Dupilumab 300 mg QW + TCS
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/107 | 0/110
Serious Adverse Events (participants affected / at risk) | 2/108 | 2/107 | 3/110
Other Adverse Events (participants affected / at risk) | 45/108 | 54/107 | 51/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo QW + TCS (N=108) | Dupilumab 300 mg Q2W + TCS (N=107) | Dupilumab 300 mg QW + TCS (N=110)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo QW + TCS (N=108) | Dupilumab 300 mg Q2W + TCS (N=107) | Dupilumab 300 mg QW + TCS (N=110)
Conjunctivitis allergic (Eye disorders) | 7 (9) | 16 (18) | 10 (11)
Conjunctivitis (Infections and infestations) | 4 (4) | 12 (14) | 8 (8)
Nasopharyngitis (Infections and infestations) | 18 (26) | 22 (29) | 18 (24)
Headache (Nervous system disorders) | 10 (17) | 10 (20) | 11 (13)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 7 (8) | 4 (7)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 18 (26) | 8 (10) | 10 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.